CLINICAL TRIAL: NCT01798238
Title: A Phase III Double-blind, Parallel Group, Randomized, Placebo-controlled Clinical Trial to Study the Efficacy and Safety of MP-513 Monotherapy in Patients With Type 2 Diabetes Mellitus
Brief Title: Teneligliptin(MP-513) Versus Placebo in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP_C302
Record Dates: First submitted 2013-02-18; First posted 2013-02-25 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus / Dipeptidyl peptidase-IV inhibitors
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo
- MP-513 group (Experimental)
  Interventions: Drug: MP-513

INTERVENTIONS:
Drug: MP-513 — form : Pink film-coated tablet for oral administration Dosage : 20mg/tablet frequency and duration: 1 tablet/day
  Arms: MP-513 group
Drug: Placebo — Pink film-coated tablet for oral administration, frequency and duration: 1 tablet/day
  Arms: Placebo group

SUMMARY:
The study design of this trial is double blind, parallel-group, randomized, placebo controlled study

DETAILED DESCRIPTION:
* Although many different oral antidiabetic agents are currently available, approximately 50% of treated Type 2 diabetic subjects do not reach currently accepted goals for HbA1c(Oral communication, American Diabetic Association, 2008)Subjects are frequently prescribed agents which can cause hypoglycemia, and/or weight gain.
* In many countries, the most commonly prescribed primary oral diabetes drug that does not cause hypoglycemia or weight gain, is metformin, but metformin can cause gastrointestinal adverse drug reactions, nausea, vomiting, diarrhea, abdominal pain and loss of appetite and other symptoms, and rare but life-threatening lactic acidosis.
* This decrease in the Power of Hydrogen Ions of the blood (<7.25) and the increase in blood lactate (> 5 mmol / L) is associated with a reduced kidney failure and if there is kidney impairment, decreased metformin clearance and thus accumulated metformin may occur lactic acidosis more frequently. Also there is inconvenience, such as adjusting metformin dose depending on patient's condition.
* MP-513 is expected to be safely used as a treatment for type 2 diabetes because it has no risk of hypoglycemia and/or weight gain which are reported in pre-existing diabetes therapies and no inconvenience related to dose adjustment depending on patient's condition, and no cases of fatal side effects.
* Furthermore the inhibitory effect on Dipeptidyl peptidase-IV was stronger and half-life was longer compared with other dipeptidyl peptidase-IV inhibitors in non-clinical trial, and blood glucose moderating effects are proven to be clinically significant in clinical trials conducted in Europe and Japan in that its development as a therapeutic agent for patients with type 2 diabetes is considered to be promising.
* Based on these previous studies, the objective of this study is to investigate the efficacy and safety in subjects with type 2 diabetes mellitus that is not adequately controlled with exercise and diet.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is aged ≥18 years at signature of the informed consent form
2. The subject has a documented diagnosis of Type 2 diabetes
3. The subject's HbA1c is 7.0%≤HbA1c<10.0% at screening visit and run-in visit
4. The subject's BMI is 20.0≤BMI≤40.0kg/m2
5. The subject's fasting plasma glucose is <15 mmol/L (270 mg/dL)at screening visit and run-in visit
6. The subject conducts a proper diet and exercise therapy for diabetes and its contents have not been changed for at least 8 week(56 days) at run-in visit(this does not apply to a subject with complications as as result of that exercise therapy is impossible)
7. The subject has not used other diabetic medicine for at least 8 week(56 days) at run-in visit
8. The subject is capable of giving informed consent, complying with the restrictions and requirements of the protocol

Exclusion Criteria:

1. The subject has a history of Type 1 diabetes or a secondary form of diabetes(Diabetes caused by the pancreatic diseases, such as chronic pancreatitis, pancreatic cancer, hemochromatosis or the overproduction of hormones antagonistic to insulin, Cushing's syndrome, Basedow's disease, pheochromocytoma, drug, insulin receptor abnormalities)
2. The subject has a history of MP-513 treatment
3. The subject has a history of habitual and excessive alcohol abuse or drug abuse, or concerns
4. The subject has a medical history of unstable angina, or heart failure(New York Heart Association class Ⅲ-IV) or any clinically significant ECG abnormalities such as ventricular tachycardia or a medical history of ventricular tachycardia
5. The subject has participated in any other clinical study involving administration of an unlicensed medicinal product within 12 weeks prior to the screening visit or is participating any other clinical study
6. The subject has received insulin within 12 months prior to the screening visit, with the exception of insulin therapy during hospitalization, insulin therapy for medical conditions not requiring hospitalization (<2 weeks duration) or use in gestational diabetes
7. Female subjects whose pregnancy test is positive or who are pregnant, lactating, or are planning to become pregnant during the study
8. The subject has serum creatinine >1.5 mg/dL(male) or >1.4 mg/dL(female)
9. The subject has aspartate-amino-transferase (AST) and alanine-amino-transferase (ALT) >2.5 times the upper limit of normal (ULN)
10. The subject has diastolic blood pressure >100 mmHg and/or systolic blood pressure >180 mmHg
11. The presence of any other condition that leads the investigator to conclude that the patient is inappropriate for inclusion in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin | Visit 1(Baseline Visit) vs Visit 7(week 24)

SECONDARY OUTCOMES:
Mean fasting plasma glucose | Visit 1(Baseline Visit) vs Visit 7(week 24)
Weight | Visit 1(Baseline Visit) vs Visit 7(week 24)
Glycosylated hemoglobin <7.0% subject percent | Visit 1(Baseline Visit) vs Visit 7(week 24)
Triglycerides | Visit 1(Baseline Visit) vs Visit 7(week 24)
Homeostatic model assessment of insulin Resistance | Visit 1(Baseline Visit) vs Visit 7(week 24)
Body mass index | Visit 1(Baseline Visit) vs Visit 7(week 24)
Low Density Lipoprotein | Visit 1(Baseline Visit) vs Visit 7(week 24)
High Density Lipoprotein | Visit 1(Baseline Visit) vs Visit 7(week 24)
Cholesterol | Visit 1(Baseline Visit) vs Visit 7(week 24)
Connecting peptide | Visit 1(Baseline Visit) vs Visit 7(week 24)
Insulin | Visit 1(Baseline Visit) vs Visit 7(week 24)
Homeostatic model assessment of beta-cell function | Visit 1(Baseline Visit) vs Visit 7(week 24)
Glycosylated hemoglobin <6.5% subject percent | Visit 1(Baseline Visit) vs Visit 7(week 24)

CONTACTS AND LOCATIONS:
Overall Officials: Sungwoo Park, Principal Investigator — Kangbuk Samsung Hospital
Locations (2):
- South Korea (2):
  - Handok INC, Seoul, Gangnam-Gu
  - Handok Pharmaceuticals CO. LTD, Seoul